CLINICAL TRIAL: NCT05380141
Title: Art and Movement at the Service of Children Who Are Victims of School Bullying
Acronym: MOUV'ON
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220339; 2022-A00430-43 (Other: ID-RCB Number)
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2023-01

CONDITIONS: Unexplained Chronic Pain; School Bullying
Keywords: Unexplained chronic pain; School bullying; Art of movement workshop; Creative art workshop; Self-esteem; Feeling of pain; Social skills
MeSH Terms: conditions — Social Skills

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients, children and adolescents referred to the chronic pain consultation of Necker Hospital with identification of school absenteeism or dropping out and having been the victim of school bullying.
  Interventions: Behavioral: Individual patient interviews

INTERVENTIONS:
Behavioral: Individual patient interviews — Two individual interviews, of one hour duration, will take place for each patient before the beginning of participating to the workshops and in the month following the end of the workshops.
  They will be led by a psychologist and a nurse from the functional pain and palliative medicine unit of Necker Hospital and 3 questionnaires will be completed during each interview.

SUMMARY:
In the context of the care of children or adolescents with unexplained chronic pain, it is not uncommon to find that some patients confide in past or present school bullying.

School bullying can have devastating consequences. Often taboo or not taken into account, it can lead to school phobia with dropout, extreme moral suffering or even reactive physical disorders. Loss of confidence, withdrawal into oneself can develop major depressive syndromes that can lead to suicidal thoughts and acting out.

The Mouv'on project offers these children/adolescents the opportunity to experience the art of movement, on the border between martial arts and dance (group sessions) and creative art (production of a street-art fresco) in order to regain confidence, restore the link to the other, discover or re-discover the relationship to the body.

It is indeed a parenthesis of relaxation, movement, breathing and meeting. The meeting of the child with himself but also with a group.

The objectives of the study are to assess the benefits of the workshops offered to children and adolescents on self-esteem and on the feeling of pain and the impact of pain on daily behavior.

DETAILED DESCRIPTION:
The pain medicine consultation at Necker Enfants Malades Hospital sees very regularly and more and more frequently children and adolescents referred for unexplained chronic pain (abdominal pain, headache, limb pain) often associated with sleep disorders, eating disorders and behavioral disorders.

Sometimes, these disorders are so important that they invade the daily life of the child and lead to school absenteeism that can go as far as dropping out of school.

It is by dint of a specific listening, of patience, of taking into account the word of the child in consultation, that often, bonds are woven and the young patients confide on the past or present school bullying.

The pain medicine consultation at Necker Enfants Malades Hospital will offer these patients the opportunity to participate in two workshop sessions:

1. st workshop: The art of movement - 10 sessions (1 hour per session) The first thing children/teenagers will discover is the importance of breathing. They will be able to reclaim it and then experiment with it in pairs, with others, in different conditions.

   This work, accompanied by an experienced teacher, will consist of connecting/reconnecting to one's body through situations involving the physique and the small and large muscle groups, gently, at each person's pace.

   Young people will learn to be in movement (martial arts / dance) and to have the right posture with regard to different situations. Thus, they will experience this connection to themselves, to the other, to others, in conditions of cooperation or conditions known as opposition.
2. nd workshop: creative art - 8 sessions (from 1 to 2 hours per session) The street-art sessions will take place in two stages. The first is the preparation phase (3 sessions) during which the participants will choose the theme and patterns.

The second stage will be the realisation phase of the mural on a wall of the Necker hospital.

This creative art will allow children and adolescents to experiment together, create, help each other, talk to each other to be able to move forward again.

These street-art sessions (art that attracts, fascinates, and is an integral part of contemporary art), could make it possible to convey ideas, values, emotions and ultimately to convey strong messages.

The creation in team will help children and adolescents to develop many social skills, such as patience, empathy, communication, respect for others, compromise, cohesion and tolerance. It will also help them develop trust in themselves and in each other.

The objectives of the study are to assess the benefits of the workshops offered to children and adolescents on self-esteem and on the feeling of pain and the impact of pain on daily behavior.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to a chronic pain consultation at the Necker hospital with identification of school absenteeism or dropping out and having been the victim of school harassment
* Non-opposition of the holders of parental authority and of the child / adolescent
* Mobility to participate in workshops
* Patients fluent in French

Exclusion Criteria:

* Patients with proven psychiatric history, unwilling to work in a group
* Patients with reduced mobility

Ages: 6 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Patients referred to a chronic pain consultation at the Necker hospital with identification of school absenteeism or dropping out and having been the victim of school harassment.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Assessment of self-esteem | 6 months
  We will use the Coopersmith Self-Esteem Inventory (CSEI), a self-administered questionnaire designed to measure attitudes toward the self in a variety of areas for children and adolescents. The CSEI consists of 58 items and yields an overall score and four separate scores representing specific aspects of self-esteem, namely, general self, social self-peers, home parents, and school academic. A set of eight additional items constitutes a lie scale. Each item is worth 2 points, making possible total scores range from 0 - 100, with higher scores relating to higher self-esteem. This questionnaire will be completed during the two individual interviews of the patient, before and 1 month after the workshops, in order to assess the benefits of workshops on self-esteem. Success will be defined for an average increase in score of 10% at the end of the workshops.

SECONDARY OUTCOMES:
Felt painful | 6 months
  The pain measurement tool will be adapted according to the age of the patient:
  * Between 6 and 10 years old: corporal diagram which will give access to both the location and the intensity of the pain, supplemented by a few questions to assess the duration, rhythm, etc.
  * From 11 years old: pain rating using a numerical scale supplemented by a few questions to assess the duration, rhythm, etc.
  This assessment will be done during the two individual interviews of the patient, before the beginning of the workshops and in the month following the end of the workshops, in order to assess the benefits of workshops offered to children and adolescents on felt painful.
  Success will be define by a loss of 2 points in average on the pain scale (0 no pain to 10 worst pain) after the workshops.
Impact of pain on daily behavior (BPI) | 6 months
  The Brief Pain Inventory (BPI) is a self-administered questionnaire use for chronic pain conditions. It is a nine items form which will give two main scores: a pain severity and a pain interference. The pain severity score is calculated from the four items about pain intensity rated from 0, no pain, to 10, pain as bad as you can imagine. The pain interference score corresponds to seven sub-items rated from 0, does not interfere, to 10, completely interferes. This questionnaire will be completed during the two individual interviews of the patient, before and 1 month after the workshops, in order to assess the benefits of workshops on the impact of pain on daily behavior. Success will be defined for an average decrease in score of 10% at the end of the workshops.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Zellner, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Céline Greco, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France